CLINICAL TRIAL: NCT05919992
Title: The Role of Glucocorticoids to Maintain Energy Homeostasis During Starvation
Brief Title: The Role of Glucocorticoids to Maintain Energy Homeostasis During Starvation (Gluco-Starve)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eleonora Seelig (Other)
Responsible Party: Sponsor-Investigator, Eleonora Seelig, Principal Investigator, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: EKNZ 2022-01837
Record Dates: First submitted 2023-03-03; First posted 2023-06-27 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Glucocorticoid Effect
Keywords: cortisol; glucocorticoids; starvation; caloric restriction; fasting
MeSH Terms: conditions — Starvation; Fasting | interventions — Metyrapone; Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled cross-over study
Who Masked: Participant, Investigator
Masking Description: Placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metyrapone And Hydrocortisone (Experimental): During one of the study periods, subjects receive hydrocortisone 19.9 mg/d subcutaneously via a pump in a pulsed fashion (eight times/day) and metyrapone per os (starting with a dose of 500 mg/d, then the dose will be increased the next days until 3000mg/d is achieved).
  Interventions: Drug: Metyrapone 250 mg Oral Tablets; Drug: Hydrocortisone 19.9mg s.c., pulsatile with a flow rate of 10μl/s
- Placebo (Placebo Comparator): During the other study period, subjects receive placebo (0,9% NaCl solution) 19.9 mg/d subcutaneously via a pump in a pulsed fashion and the same dose of placebo tablets p.o instead of metyrapone
  Interventions: Drug: Placebo 250 mg Tablets; Drug: Placebo (0,9% NaCl solution)

INTERVENTIONS:
Drug: Metyrapone 250 mg Oral Tablets — During one phase of the study: Metyrapone (pills of 250mg) on empty stomach: Day 1 0-1-1, day 2 1-2-2, day 3 2-3-3 day 4 3-4-4 day 5 4-4-4 day 6 4-4-4 day 7 4-0-0
  Arms: Metyrapone And Hydrocortisone
Drug: Hydrocortisone 19.9mg s.c., pulsatile with a flow rate of 10μl/s — Hydrocortisone will be delivered subcutaneously via a pump in a pulsed fashion with a flow rate of 10μl/s from day 1 to day 7 in a total daily dose of 19.9mg
  Arms: Metyrapone And Hydrocortisone
Drug: Placebo 250 mg Tablets — During another phase of the study: identical looking placebo pills starting Day 1 0-1-1, day 2 1-2-2, day 3 2-3-3 day 4 3-4-4 day 5 4-4-4 day 6 4-4-4 day 7 4-0-0
  Arms: Placebo
Drug: Placebo (0,9% NaCl solution) — Placebo (0,9% NaCl solution) 19.9 mg/d subcutaneously via a pump in a pulsed fashion with a flow rate of 10μl/s from day 1 to day 7
  Arms: Placebo

SUMMARY:
In a randomized, cross-over study, 20 healthy volunteers will receive a block and replace therapy that mimics physiological GC rhythm (metyrapone plus hydrocortisone) or placebo. Participants will undergo two identical fasting periods with each treatment. With the block and replace therapy, fasting-induced GC peak will be suppressed. Metabolic and autonomic parameters will be compared to reveal whether GCs mediate the physiological adaptions to caloric restriction.

Understanding acute effects of GCs upon caloric restriction is critical, since repetitive disruptions of GC secretion may become harmful in chronic conditions.

DETAILED DESCRIPTION:
Obesity is one of the major causes of morbidity and mortality worldwide. Achieving long-term weight loss is challenging, as the body counteracts weight loss to preserve energy by increasing appetite and lowering energy expenditure. These physiological defense mechanisms are the main obstacle to successful weight reduction in obese people.

Therefore, identifying the signals that defend body weight during caloric restriction is essential for developing new antiobesity drugs. Corticosteroids mediate the physiological defense to starvation in rodents. Whether cortisol has the same impact on humans is unknown.

Therefore, we investigate whether cortisol regulates the physiological adaptions to caloric restriction in humans.

The general objective of this project is to investigate whether cortisol mediates physiological adaptions to caloric restriction.

The primary objective is to test whether cortisol mediates the increased appetite during caloric restriction.

Secondary objectives are to test whether the cortisol response to caloric restriction affects satiation, satiety, energy expenditure, substrate utilization, blood pressure, weight, body composition, secretion of neuroendocrine hormones, lipids, glucose, ketone bodies, sympathetic nervous system activity, immune cells, and inflammatory markers.

This is a double-blind, randomized, placebo-controlled crossover study.

After screening, subjects will be randomized to two crossover 7-day study periods with a wash-out period of 28 days:

A) Participants will receive hydrocortisone 19.9 mg/d subcutaneously via a pump in a pulsed fashion (eight times/day) and metyrapone capsules per os (starting with a dose of 500 mg/d on day 1 to 3000mg/d on day 5, and then will be kept constant until day 7).

B) Participants will receive a placebo (0,9% NaCl solution) subcutaneously via a pump in a pulsed fashion and identical-looking placebo capsules per os with the same regimen as for metyrapone.

During both study periods, participants will undergo two days of caloric restriction.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 - 27 kg/m2
* Weight stability for 6 months prior to the trial (+/- 2kg)

Exclusion Criteria:

* Previous medical history for any chronic condition in the last three months, active disease or abnormal physical examination as verified by a qualified physician.
* Casual smoking (>6 cigarettes per day)
* Frequent, heavy alcohol consumption (>30g/day)
* Frequent, heavy caffeine consumption (>4 caffeinated drinks/day)
* Regular physical exercise (>4hrs per week)
* Shift workers
* Participation in an investigational drug trial within the past two months
* Intake of any drugs (prescribed, over the counter or recreational), within 48 hours of the study initiation
* Intake of any steroids (including topical or inhaler) six month prior to the study
* Known allergy to metyrapone or hydrocortisone
* Inability or unwillingness to provide informed consent

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Satiation | Two 7-day intervention periods
  Amount of food intake with ad libitum buffet

SECONDARY OUTCOMES:
Satiety | Two 7-day intervention periods
  Appetite rating by visual analog scale, minimum value 0, maximum value 100
Food preference | Two 7-day intervention periods
  Amount of fat/ protein/carbohydrates consumed during ad libitum buffet
Energy expenditure | Two 7-day intervention periods
  Basal metabolic rate, diet-induced thermogenesis
Substrate utilization | Two 7-day intervention periods
  Respiratory quotient
Blood pressure | Two 7-day intervention periods
  Blood pressure
Weight | Two 7-day intervention periods
  Body weight
Body composition | Two 7-day intervention periods
  measured with DEXA-Scans and body impedance analysis
Neuroendocrine hormones | Two 7-day intervention periods
  Leptin, thyroid hormones, insulin, c-peptide, growth hormone, IGF1, catecholamines, GLP-1, GIP, glucagon, PYY, CCK, ghrelin, GDF-15, cortisol total and free, ACTH, renin, aldosterone, pregnenolone, progesterone, 11-deoxycorticosterone, corticosterone, 18-hydroxycorticosterone, 17-hydroxypregnenolone, 17-hydroxyprogesterone, 11-deoxycortisol, oxytocin, FGF-21
Lipids | Two 7-day intervention periods
  Total cholesterol, LDL-cholesterol, HDL-cholesterol, and triglycerides
Glucose | Two 7-day intervention periods
  measured via blood sample
Insulin sensitivity | Two 7-day intervention periods
  measured via blood sample
Ketone bodies | Two 7-day intervention periods
  measured via blood sample
Sympathetic nervous system activity | Two 7-day intervention periods
  measured via ECG: Heart rate, interbeat interval, high-frequency activity, low-frequency activity, root mean square of successive differences
Immune cells | Two 7-day intervention periods
  Peripheral blood mononuclear cells (PBMCs)
Inflammatory markers | Two 7-day intervention periods
  IL-6, IL-1RA, IL-8, CRP
Motivation to eat | Two 7-day intervention periods
  clicking speed computer test
Pleasure from eating | Two 7-day intervention periods
  Fonts rating test
Measure of behavioural approach and behavioural inhibition system | Two 7-day intervention periods
  Questionnaire
Eating behaviour type | Two 7-day intervention periods
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No